CLINICAL TRIAL: NCT07115576
Title: Radiofrequency Ablation for the Treatment of Benign Thyroid Nodules: A Prospective Study
Acronym: RFAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hue University of Medicine and Pharmacy (Other)
Collaborators: Da Nang Family General Hospital (Other)
Responsible Party: Principal Investigator, Le Van Chi, professor, Hue University of Medicine and Pharmacy
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H2023/050
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Benign Thyroid Nodules
Keywords: Benign thyroid nodules; Radiofrequency Ablation; Prospective Study
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- primary end-point (Experimental): To evaluate the efficacy of RFA procedure in reducing the volume of benign cystic thyroid nodules, measured by the volume reduction rate (VRR) at 1, 6, and 12 months post-procedure.
  Interventions: Procedure: Radiofrequency ablation alone
- Secondary end-point (Experimental): • To assess the safety of RFA procedure, including the incidence of major and minor complications.
  Interventions: Procedure: Radiofrequency ablation alone

INTERVENTIONS:
Procedure: Radiofrequency ablation alone — Radiofrequency ablation (RFA) is a minimally invasive procedure used to treat benign thyroid nodules without surgery. It involves inserting a thin, needle-like electrode into the nodule under ultrasound guidance. Using high-frequency alternating current, the electrode generates heat to destroy targeted thyroid tissue, causing the nodule to shrink over time.
  Other Names: RFA

SUMMARY:
Title:

Radiofrequency Ablation for the Treatment of Benign Thyroid Nodules: A Prospective Study

Purpose:

The goal of this clinical trial is to learn if single-session radiofrequency ablation (RFA) can effectively reduce the volume of benign thyroid nodules in adults. It will also evaluate the safety of the RFA procedure.

The main questions it aims to answer are:

1. Does RFA procedure reduce the size of thyroid nodules (measured by volume reduction rate - VRR)?
2. What medical problems or complications do participants experience after undergoing RFA?
3. How does RFA affect thyroid hormone levels (TSH, FT4)?
4. Is RFA equally effective in purely cystic nodules, solid nodules, and predominantly cystic nodules?

Comparator:

This is a single-arm study, so there is no placebo or comparison treatment group. All participants will undergo RFA, and the results will be assessed over time.

Participants will:

* Undergo one session of RFA for benign thyroid nodules.
* Be followed up with clinical visits and ultrasound assessments at 1, 6, and 12 months.
* Have thyroid hormone levels tested and nodule size measured by ultrasound at each follow-up.
* Be monitored for any side effects or complications such as voice changes, pain, or bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thyroid nodules, confirmed by ultrasound.
* Presence of compressive symptoms (e.g., dysphagia, neck pressure) or cosmetic concerns.
* Documented thyroid function tests (serum free thyroxine [FT4] and thyrotropin [TSH]).
* Cytology-confirmed benign thyroid nodules via one or two ultrasound-guided fine-needle aspiration (FNA) procedures.
* Refusal of surgical treatment.
* Ability to complete follow-up assessments at 1, 6, and 12 months post-procedure.

Exclusion Criteria:

* Malignant or indeterminate cytology on FNA.
* Contraindications to RFA (e.g., severe coagulopathy, pregnancy).
* Uncontrolled thyroid dysfunction (e.g., hyperthyroidism or hypothyroidism).
* Inability to provide informed consent or comply with follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Volume Reduction Rate (VRR) | 1 month; 6 months; 12 months
  The volume reduction rate (VRR) is used to assess the effectiveness of radiofrequency ablation (RFA) in shrinking thyroid nodules over time. It is calculated as the percentage decrease in nodule volume compared to baseline:
  VRR (%) = [(Initial Volume - Follow-up Volume) / Initial Volume] × 100
  In this study, VRR will be measured at 1, 6, and 12 months after the RFA procedure using ultrasound. A VRR greater than 50% is generally considered a successful therapeutic outcome. Tracking VRR at these time points helps evaluate the progressive reduction in nodule size and the long-term efficacy of the treatment.
volume reduction rate (VRR) at 1, 6, and 12 months post-procedure. | 1 month; 6 months; 12 months
  The volume reduction rate (VRR) is used to assess the effectiveness of radiofrequency ablation (RFA) in shrinking thyroid nodules over time. It is calculated as the percentage decrease in nodule volume compared to baseline:
  VRR (%) = [(Initial Volume - Follow-up Volume) / Initial Volume] × 100
  In this study, VRR will be measured at 1, 6, and 12 months after the RFA procedure using ultrasound. A VRR greater than 50% is generally considered a successful therapeutic outcome. Tracking VRR at these time points helps evaluate the progressive reduction in nodule size and the long-term efficacy of the treatment.

SECONDARY OUTCOMES:
Assess the safety of single-session RFA | 1 month, 6 months, 12 months
  The safety of radiofrequency ablation (RFA) procedure for benign thyroid nodules is evaluated by monitoring the incidence and severity of complications following the procedure. Complications are classified as major (e.g., permanent voice changes, significant bleeding requiring intervention, hospitalization) or minor (e.g., transient pain, temporary voice hoarseness, mild swelling).
  All adverse events are recorded during and after the procedure, and at follow-up visits at 1, 6, and 12 months. Safety assessments follow international guidelines for image-guided tumor ablation. The absence of serious complications and a low rate of minor, self-limiting events indicate that single-session RFA is a safe and well-tolerated alternative to surgery for selected patients with benign thyroid nodules.

CONTACTS AND LOCATIONS:
Locations (1):
- Hue University of Medicine and Pharmacy, Hue University,, Huế, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen VB, Le TB, Van CL. Single-session radiofrequency ablation for the treatment of benign cystic thyroid nodules: A prospective study. PLoS One. 2026 Feb 4;21(2):e0341556. doi: 10.1371/journal.pone.0341556. eCollection 2026. PMID 41637422

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT07115576/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: study protocol and Statistical Analysis Plan version 2 (2025-12-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT07115576/Prot_SAP_002.pdf